CLINICAL TRIAL: NCT06572033
Title: Transference of Established Simulated Skills (TEST) Trial: Tracking Transference of Positive Pressure Ventilation Skills From Simulation to Delivery Room.
Brief Title: Transference of Established Simulated Skills (TEST) Trial
Acronym: TEST
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Vishal Kapadia, Associate Professor at UT Southwestern, University of Texas Southwestern Medical Center
Other Study IDs: STU 2023-1099
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Respiratory Distress
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Respiratory Therapists: This cohort consists of respiratory therapists (RTs) who are actively involved in both simulation-based training sessions and actual neonatal deliveries. Participants will have varying levels of experience, from newly qualified to seasoned professionals. During the study, RTs will perform positive pressure ventilation (PPV) on both neonatal mannequins in the simulation lab and on newborns in the delivery room. Their performance will be measured using a respiratory function monitor (RFM), focusing on parameters such as mask leak, peak inspiratory pressure (PIP), positive end-expiratory pressure (PEEP), and exhaled tidal volume (eVT). The goal is to assess the transferability of their skills from simulation to real-life scenarios.
  Interventions: Behavioral: Simulation
- Newborn Infants: This cohort consists of respiratory therapists (RTs) who are actively involved in both simulation-based training sessions and actual neonatal deliveries. Participants will have varying levels of experience, from newly qualified to seasoned professionals. During the study, RTs will perform positive pressure ventilation (PPV) on both neonatal mannequins in the simulation lab and on newborns in the delivery room. Their performance will be measured using a respiratory function monitor (RFM), focusing on parameters such as mask leak, peak inspiratory pressure (PIP), positive end-expiratory pressure (PEEP), and exhaled tidal volume (eVT). The goal is to assess the transferability of their skills from simulation to real-life scenarios.

INTERVENTIONS:
Behavioral: Simulation — Observational study with simulations.
  Groups: Respiratory Therapists

SUMMARY:
This study aims to determine if skills learned in the simulation lab, specifically in managing mask leak during positive pressure ventilation (PPV), translate effectively to the delivery room. By comparing the performance of healthcare providers on mannequins in the lab to their performance on newborns in the delivery room, the study seeks to establish a Ventilation Performance Score (VPS) based on data from a respiratory function monitor. The primary hypothesis is that a provider's ability to minimize mask leak on a mannequin correlates with their ability to do so with a newborn. The prospective observational TEST Trial will use the Monivent Neo100 to collect and analyze PPV data, comparing key parameters like mask leak and VQS between the two settings to assess correlations. Secondary analysis will explore individual aspects of PPV, such as PIP, PEEP, and eVT.

DETAILED DESCRIPTION:
Objectives: The aim of this study is to establish evidence that supports the transfer of skills learned in the simulation lab to the delivery room. The objective of this study is to compare the performance of positive pressure ventilation (PPV) in the simulation lab to the performance of the same individual in the delivery room. Our goal is to establish a comparison between parameters measured on the simulator and those obtained from real newborn infants, specifically looking at mask leak. Our approach hopes to develop a ventilation performance score (VPS) in the process that will be based on objective data collected using a respiratory function monitor (RFM). The primary hypothesis is that the quality of a qualified provider's ability to circumvent mask leak on a mannequin correlates with the ability of the same provider to circumvent mask leak observed on a newborn infant.

Design and outcomes: TEST Trial is a prospective observational study to assess differences in the participants ability to avoid mask leak while performing PPV and in the process allow the investigators to develop a ventilatory performance score in the simulation lab and the delivery room. We will use the RFM Monivent Neo100 to gather PPV data in both the simulation lab from the mannequins and newborns in the delivery room. The study will compare mask leak as well as VPS in the simulation room to mask leak and VPS in the delivery room to assess for correlations. In addition, the investigators will conduct secondary analysis on each individual domain of positive pressure ventilation, such as PIP, PEEP, eVT, etc.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Respiratory Therapists (RTs)

Inclusion Criteria:

* Respiratory Therapists who are employed in the Neonatal Intensive Care Unit (NICU) at Parkland Hospital.
* RTs who actively participate in neonatal deliveries.

Exclusion Criteria:

* Respiratory Therapists classified as "float" RTs, meaning those who do not have a permanent assignment in the NICU.
* RTs who intend to leave the institution within the upcoming year.

Inclusion and Exclusion Criteria for Newborn Infants

Inclusion Criteria:

* Newborn infants who require positive pressure ventilation (PPV) immediately after birth in the delivery room.
* Infants of various gestational ages and birth weights, representing a broad spectrum of neonatal resuscitation scenarios.

Exclusion Criteria:

* Newborns who do not require PPV after birth.
* Infants for whom the use of the respiratory function monitor (RFM) is not feasible due to medical or technical reasons.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Respiratory Therapists (RTs):
     Demographics: This group includes Respiratory Therapists employed in the Neonatal Intensive Care Unit (NICU) at Parkland Hospital. Participants have varying levels of experience, ranging from newly certified RTs to those with extensive experience in neonatal care.
  2. Newborn Infants:
  Demographics: This group includes newborn infants requiring positive pressure ventilation (PPV) immediately after birth in the delivery room. Infants included in the study will vary in gestational age, birth weight, and clinical condition, representing a broad range of neonatal resuscitation scenarios.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Correlation of mask leak performance | 1 year
  Correlation between the percentage of mask leak observed during positive pressure ventilation (PPV) on a mannequin in the simulation laboratory and the percentage of mask leak observed during PPV on a newborn infant in the delivery room.

SECONDARY OUTCOMES:
Correlation of Ventilation Performance Score (VPS) | 1 year
  Correlation of Ventilation Performance Score (VPS) between the simulation lab and the delivery room.
Correlation of submetrics of VPS | 1 year
  Correlation of submetrics of VPS (such as TVe, mask seal, PIP, PEEP, etc.) between the simulation lab and the delivery room.

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided